CLINICAL TRIAL: NCT04198285
Title: Post-Operative Voiding After Gynecological Surgery (POVAGS) Trial: a Randomized Controlled Trial on Retrograde Bladder Filling After Outpatient Gynaecological Laparoscopy
Brief Title: Post-Operative Voiding After Gynecological Surgery Trial
Acronym: POVAGS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to cancellation of elective surgery (Covid-19)
Sponsor: Women's College Hospital (Other)
Responsible Party: Principal Investigator, Jonathon Solnik, Site Chief of Gynecology, Women's College Hospital
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Other
Other Study IDs: 2019-0110-E
Record Dates: First submitted 2019-12-12; First posted 2019-12-13 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Urinary Retention; Postoperative Complications; Surgery
Keywords: laparoscopy, urinary retention
MeSH Terms: conditions — Urinary Retention; Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retrograde filled (Experimental): This arm will contain patients who had retrograde bladder filling upon completion of surgery with 200 milliliters (mL) of sterile saline.
  Interventions: Procedure: Retrograde bladder filling
- Control (No Intervention): This arm will contain patients who simply had the urinary catheter removed upon completion of surgery, and were left with an empty bladder.

INTERVENTIONS:
Procedure: Retrograde bladder filling — The bladder will be filled with a large syringe through the urinary catheter (which is left in place for the surgery) with 200mL of sterile saline, and then the catheter will be removed.
  Arms: Retrograde filled

SUMMARY:
To determine whether partially filling the bladder after outpatient gynaecological laparoscopy expedites time to first void and discharge. Methods: A single site, single-blinded, randomized control trial in which eligible patients undergo partial retrograde bladder filling immediately post-operatively compared to bladder drainage and foley catheter removal. Primary outcome is time to first void, secondary outcomes include time to discharge, post-operative complications and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Undergoing elective laparoscopy for a gynaecological indication
* Plan for same day discharge
* Able to provide informed consent

Exclusion Criteria:

* Pregnancy
* Undergoing procedure for pelvic organ prolapse, stress urinary incontinence, or nerve detrapment
* Prior hysterectomy, or incontinence/pelvic organ prolapse procedures
* Pre-existing voiding dysfunction
* Known recurrent urinary tract infections
* Known genito-urinary malformations
* Known for neuromuscular disorders such as multiple sclerosis
* Use of anticholinergic medication
* Intraoperative bladder related complications
* Need for discharge with indwelling foley catheter
* Patients requiring overnight admission for any reason

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — patients undergoing gynecological surgery
Enrollment: 42 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-04-27 (Actual)

PRIMARY OUTCOMES:
Time to first void | 3 hours
  Time in minutes from arrival in post-operative anesthesia unit (PACU) to first void

SECONDARY OUTCOMES:
Time to discharge | 8 hours
  Time in minutes from arrival in PACU to discharge from PACU
Post-operative complications | 1 week following surgery
  Urinary tract infections, or other reported complications
Patient satisfaction | 1 week
  Patients' subjective experience in both groups regarding time spent in PACU and first postoperative week
Post-operative pain | Assessed at the 1 hour mark
  visual analogue scale of postoperative pain, assessed in PACU

CONTACTS AND LOCATIONS:
Overall Officials: Ally Murji, MD, Principal Investigator — Women's College Hospital
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moawad G, Tyan P, Marfori C, Abi Khalil E, Park D. Effect of postoperative partial bladder filling after minimally invasive hysterectomy on postanesthesia care unit discharge and cost: a single-blinded, randomized controlled trial. Am J Obstet Gynecol. 2019 Apr;220(4):367.e1-367.e7. doi: 10.1016/j.ajog.2018.12.034. Epub 2019 Jan 9. PMID 30639089
- [Derived] Zakhari A, Paek W, Chan W, Edwards D, Matelski J, Solnik MJ, Murji A. Retrograde Bladder Filling after Laparoscopic Gynecologic Surgery: A Double-blind Randomized Controlled Trial. J Minim Invasive Gynecol. 2021 May;28(5):1006-1012.e1. doi: 10.1016/j.jmig.2020.09.019. Epub 2020 Oct 3. PMID 33017685